CLINICAL TRIAL: NCT05193370
Title: A Randomized Controlled Pilot Trial of Angiotensin II Versus Vasopressin as Second-line Vasopressor in the Treatment of Septic Shock
Brief Title: Angiotensin II vs. Vasopressin in Septic Shock
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Funding and protocol changes. Replaced with new pilot trial.
Sponsor: University of New Mexico (Other)
Collaborators: La Jolla Pharmaceutical Company (Industry); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-040; UL1TR001449 (NIH)
Record Dates: First submitted 2021-12-09; First posted 2022-01-14 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Septic Shock
Keywords: septic shock; vasopressor; angiotensin II; vasopressin; renin; randomized controlled trial
MeSH Terms: conditions — Shock, Septic; Diabetes Insipidus | interventions — Angiotensin II; Giapreza; Vasopressins; Arginine Vasopressin

STUDY DESIGN:
Intervention Model Description: single-center, open-label pragmatic randomized controlled pilot trial using block randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- angiotensin II (intervention) (Experimental): For patients randomized to the intervention group, once the dose of background norepinephrine reaches ≥0.2 mcg/kg/min for ≥30 minutes, angiotensin II will be started at a dose of 20 ng/kg/min (recommended starting dose in package insert). Thereafter, angiotensin II and norepinephrine will both be titrated according to the schema in UNM Hospitals Nursing Department Titration Guideline. Angiotensin II treatment will be capped at 72h, at which point (if a second vasopressor is still needed) the patient will be started on an alternative agent.
  Interventions: Drug: Angiotensin II
- vasopressin (standard of care) (Active Comparator): In patients randomized to the control group, once the dose of background norepinephrine reaches ≥0.2 mcg/kg/min for ≥30 minutes, vasopressin will be used at a fixed dose of 0.04 units/min and norepinephrine will be titrated per usual standard of care (as also outlined in the UNM Hospitals Nursing Department Titration Guideline).
  Interventions: Drug: Vasopressin

INTERVENTIONS:
Drug: Angiotensin II — Angiotensin II (Giapreza) is a pharmacologic version of a naturally occurring hormone of the same name, peptide hormone of the renin-angiotensin-aldosterone system (RAAS), that was FDA-approved in 2017 as a vasoconstrictive agent in the treatment of vasodilatory shock.
  Other Names: Giapreza
  Arms: angiotensin II (intervention)
Drug: Vasopressin — Vasopressin (Vasostrict) is a pharmacologic version of a naturally occurring peptide hormone that serves as a vasoconstrictive agent in the treatment of vasodilatory shock.
  Other Names: Vasostrict
  Arms: vasopressin (standard of care)

SUMMARY:
This will be a randomized controlled unblinded pragmatic single-center pilot trial of the use of vasopressin vs. angiotensin II as a second-line vasopressor in patients with septic shock and persistent hypotension despite moderate-to-high doses of norepinephrine.

DETAILED DESCRIPTION:
Sepsis affects >1 million Americans yearly and, when septic shock ensues, is associated with high morbidity and mortality. Though first-line norepinephrine is standard of care, there are limited prospective data to guide the choice of additional vasopressors in septic shock. While more studies are needed, preliminary data suggest that the vasopressor angiotensin II (AngII) may improve outcomes in septic shock.

This study is a pilot randomized controlled trial (RCT) comparing AngII (intervention) and vasopressin (standard of care) as second-line vasopressors in septic shock. The goal is to demonstrate feasibility of a large multicenter RCT and eventually to demonstrate that AngII use improves important endpoints (e.g., mortality, need for organ support) in all or certain subsets of patients with septic shock.

Furthermore, there are no biomarkers currently available and validated to guide the choice of vasopressor therapy in septic shock. In this study the investigators will investigate serum renin as such a biomarker. Renin has been shown in preliminary studies to accurately predict mortality in septic shock, outperforming lactate, and to predict beneficial response to AngII. The investigators aim to validate the use of renin as a biomarker in septic shock and prove its utility in guiding vasopressor selection, with the goal of incorporating renin levels at specified time points and/or change in renin levels into an algorithm used to select patients for AngII therapy in the subsequent large multicenter RCT.

ELIGIBILITY:
Inclusion Criteria:

* 1. Adult patients ≥18 years-old with vasodilatory shock refractory to norepinephrine monotherapy, defined as those who require ≥0.2 mcg/kg/min to maintain a MAP between 65-70 mmHg. Patients will be screened once they require ≥0.1 mcg/kg/min of norepinephrine and, if eligible, may be consented at this point. Study drug (angiotensin II or vasopressin) will be initiated once norepinephrine dose reaches ≥0.2 mcg/kg/min for at least 30 minutes.
* 2. Patients are required to have central venous and arterial catheters present, and they are expected to remain in place for at least the initial 72 hours of study.
* 3. Patients are required to have an indwelling urinary catheter present, and it is expected to remain in place for at least the 72 hours of study.
* 4. Patients must have received 20-30 mL/kg of crystalloid over the previous 24-hour period, as clinically appropriate, and no longer be fluid responsive as per UNMH protocol. By UNMH protocol, lack of fluid responsiveness is considered a failure to increase stroke volume, stroke volume index, cardiac output, or cardiac index (typically measured by non-calibrated pulse contour analysis using a FloTrac device) by at least 10% after a 500-mL crystalloid bolus or a passive leg raise. Patients for whom the treating physicians feel that 20 mL/kg of crystalloid may be clinically inappropriate can qualify for the study if the reason for withholding further IV fluids is documented.
* 5. Patient or (in patients unable to consent) legal authorized representative (LAR) is willing and able to provide written informed consent and comply with all protocol requirements.
* 6. Approval from the attending physician and clinical pharmacist conducting the study.

Exclusion Criteria:

* 1. Patients who are < 18 years of age.
* 2. Patients diagnosed with acute occlusive coronary syndrome requiring intervention and/or cardiogenic shock.
* 3. Patients with or suspected to have abdominal aortic aneurysm or aortic dissection.
* 4. Acute stroke.
* 5. Patients with acute mesenteric ischemia or those with a history of mesenteric ischemia.
* 6. Patients with known Raynaud's phenomenon, systemic sclerosis, or vasospastic disease.
* 7. Patients on veno-arterial (VA) ECMO.
* 8. Patients with liver failure with a Model for End-Stage Liver Disease (MELD) score of ≥30.
* 9. Patients with burns covering >20% of total body surface area.
* 10. Patients with a history of asthma or COPD with active acute bronchospasm or (if not mechanically ventilated) with an acute exacerbation of their asthma/COPD requiring the use of inhaled bronchodilators.
* 11. Patients requiring more than 500 mg daily of hydrocortisone or equivalent glucocorticoid medication as a standing dose.
* 12 Patients with an absolute neutrophil count (ANC) of < 1,000/mm3.
* 13. Patients with hemorrhagic shock OR active bleeding AND an anticipated need (within 48 hours of initiation of the study) for transfusion of >4 units of packed red blood cells.
* 14. Patients with active bleeding AND hemoglobin < 7g/dL or any other condition that would contraindicate serial blood sampling.
* 15. Untreated venous thromboembolism (VTE) or inability to tolerate pharmacologic VTE prophylaxis.
* 16. Patients with a known allergy to mannitol.
* 17. Patients with an expected survival of <24 hours, SOFA score ≥ 16, or death deemed to be imminent or inevitable during the admission
* 18. Either the attending physician or patient and/or substitute decision-maker are not committed to all active treatment (e.g., DNR status).
* 19. Patients who are known to be pregnant at the time of screening. [All women ≤50 years-old will need a negative serum pregnancy test (serum quantitative beta-hCG) to enroll.]
* 20. Prisoner status
* 21. Patients who are current participating in another interventional clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-03 (Estimated); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients who achieve blood pressure (BP) goal (MAP ≥65 mmHg) at 3 hours post-drug initiation | 3 hours
  The primary endpoint will be the percentage of patients who achieve BP goal, specifically mean arterial pressure (MAP) of ≥65 mmHg, at the 3-hour time point. The primary endpoint will be binary (yes/no achievement of BP goal). Failure to respond to study drug will defined as any of the following: (1) MAP <65 mmHg at 3 hours, (2) Need for increase in background norepinephrine to >0.2 mcg/kg/min despite the addition of the study drug, or (3) Need for a third vasopressor.

SECONDARY OUTCOMES:
BP goal at other time points | Up to 72 hours
  The primary endpoint will be re-assessed at multiple additional time points (1 hour, 6 hours, 12 hours, 24 hours, 48 hours, and 72 hours)
Time to shock reversal | Up to 72 hours
  Time to sustained shock reversal (vasopressor independence).
Change in catecholamine dose | Up to 72 hours
  Change in catecholamine dose (as quantified in norepinephrine equivalents) at 1 hour, 3 hours, 6 hours, 12 hours, 24 hours, 48 hours, and 72 hours.
SOFA score | Up to 72 hours
  Change in Sequential Organ Failure Assessment (SOFA) scores and/or organ-specific SOFA sub-scores at 1 hour, 3 hours, 6 hours, 12 hours, 24 hours, 48 hours, and 72 hours. SOFA ranges from 0 to 24 with higher score indicating higher illness severity.
Acute Kidney Injury (AKI) | Up to 28 days
  Frequency of AKI, as defined by KDIGO (Kidney Disease: Improving Global Outcomes) criteria.
Freedom from Renal Replacement Therapy (RRT) | Up to 28 days
  Days free from RRT (in first 28 days post study drug initiation)
Ventilator-free days | Up to 28 days
  Days free from invasive mechanical ventilation (in first 28 days post drug initiation)
ICU LOS | Though study completion, up to 1 year
  ICU length of stay
Hospital LOS | Though study completion, up to 1 year
  Hospital length of stay
ICU mortality | Up to 28 days
  ICU mortality (defined as binary yes/no, until ICU discharge or 28 days from drug initiation)
Hospital mortality | Up to 28 days
  Hospital mortality (defined as binary yes/no, until hospital discharge or 28 days from drug initiation)
Renin levels | Up to 3 hours
  Renin levels will be obtained at 4 times points: at consent/pre-baseline; at baseline/time 0 (drug initiation); 1 hour post-initiation; and 3 hours post-initiation. The investigators will also perform exploratory analyses of differences in the primary and secondary outcomes as stratified by renin levels and/or changes in renin level.
Subgroup analyses | Though study completion, up to 1 year
  The investigators will perform exploratory analyses of the other primary and secondary outcomes as stratified by disease severity (as measured by SOFA scores).
  All the other primary and secondary outcomes will be also re-analyzed to assess for differences within the following subgroups:
  * presence or absence of AKI
  * presence or absence of ARDS
Prespecified Adverse Events | Up to 28 days
  For these to be considered adverse events (AEs) they must be new hospital-acquired events which developed after randomization.
  The pre-defined AEs that will be tracked will include the rates of:
  * New venous thromboembolism (VTE) or arterial thrombosis diagnosed during hospital stay.
  * Atrial fibrillation
  * Tachycardia
  * Lactic acidosis
  * Peripheral limb/digit ischemia
  * Intestinal ischemia
  * Thrombocytopenia
  * Hyperglycemia
  * Confirmed infection (with infecting organism confirmed by culture or other identification method; administration of appropriate antibiotic therapy; and clinical documentation of infection)
  * Any other AE that is felt to be potentially related to study drug

CONTACTS AND LOCATIONS:
Overall Officials: Joao P Teixeira, MD, Principal Investigator — University of New Mexico School of Medicine; Nathan D Nielsen, MD MSc, Principal Investigator — University of New Mexico School of Medicine
Locations (1):
- University of New Mexico Health Sciences Center, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khanna A, English SW, Wang XS, Ham K, Tumlin J, Szerlip H, Busse LW, Altaweel L, Albertson TE, Mackey C, McCurdy MT, Boldt DW, Chock S, Young PJ, Krell K, Wunderink RG, Ostermann M, Murugan R, Gong MN, Panwar R, Hastbacka J, Favory R, Venkatesh B, Thompson BT, Bellomo R, Jensen J, Kroll S, Chawla LS, Tidmarsh GF, Deane AM; ATHOS-3 Investigators. Angiotensin II for the Treatment of Vasodilatory Shock. N Engl J Med. 2017 Aug 3;377(5):419-430. doi: 10.1056/NEJMoa1704154. Epub 2017 May 21. PMID 28528561
- [Background] Tumlin JA, Murugan R, Deane AM, Ostermann M, Busse LW, Ham KR, Kashani K, Szerlip HM, Prowle JR, Bihorac A, Finkel KW, Zarbock A, Forni LG, Lynch SJ, Jensen J, Kroll S, Chawla LS, Tidmarsh GF, Bellomo R; Angiotensin II for the Treatment of High-Output Shock 3 (ATHOS-3) Investigators. Outcomes in Patients with Vasodilatory Shock and Renal Replacement Therapy Treated with Intravenous Angiotensin II. Crit Care Med. 2018 Jun;46(6):949-957. doi: 10.1097/CCM.0000000000003092. PMID 29509568
- [Background] Gordon AC, Mason AJ, Thirunavukkarasu N, Perkins GD, Cecconi M, Cepkova M, Pogson DG, Aya HD, Anjum A, Frazier GJ, Santhakumaran S, Ashby D, Brett SJ; VANISH Investigators. Effect of Early Vasopressin vs Norepinephrine on Kidney Failure in Patients With Septic Shock: The VANISH Randomized Clinical Trial. JAMA. 2016 Aug 2;316(5):509-18. doi: 10.1001/jama.2016.10485. PMID 27483065
- [Background] Busse L, Albertson T, Gong M. Outcomes in patients with acute respiratory distress syndrome receiving angiotensin II for vasodilatory shock. Crit Care. 2018;22(Suppl 1):82.
- [Background] Gleeson PJ, Crippa IA, Mongkolpun W, Cavicchi FZ, Van Meerhaeghe T, Brimioulle S, Taccone FS, Vincent JL, Creteur J. Renin as a Marker of Tissue-Perfusion and Prognosis in Critically Ill Patients. Crit Care Med. 2019 Feb;47(2):152-158. doi: 10.1097/CCM.0000000000003544. PMID 30653055
- [Background] Bellomo R, Forni LG, Busse LW, McCurdy MT, Ham KR, Boldt DW, Hastbacka J, Khanna AK, Albertson TE, Tumlin J, Storey K, Handisides D, Tidmarsh GF, Chawla LS, Ostermann M. Renin and Survival in Patients Given Angiotensin II for Catecholamine-Resistant Vasodilatory Shock. A Clinical Trial. Am J Respir Crit Care Med. 2020 Nov 1;202(9):1253-1261. doi: 10.1164/rccm.201911-2172OC. PMID 32609011

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-20): https://cdn.clinicaltrials.gov/large-docs/70/NCT05193370/Prot_SAP_000.pdf
  • Informed Consent Form (2021-10-01): https://cdn.clinicaltrials.gov/large-docs/70/NCT05193370/ICF_001.pdf